CLINICAL TRIAL: NCT05008016
Title: Procalcitonin Level and the High Risk of Mortality in 30 Days , in Critically Ill Patients Infected by SARS-CoV-2, Experience of a North African Hospital University , Cases Series.
Brief Title: Procalcitonin Level and the High Risk of Mortality in 30 Days in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Patient , Cases Series.
Status: Completed | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Younes Oujidi, Principal Investigator, Mohammed VI University Hospital
Other Study IDs: Anaesthesia and Resuscitation
Record Dates: First submitted 2021-08-11; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: the Relationship Between Procalcitonin and 30-day Mortality in COVID Patients
Keywords: COVID; Procalcitonine; Mortality

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Procalcitonine analysed: The invistagatore had analysed the Procalcitonine of patient that survived and the non Survived frome COVID infection in Intensive care departement

SUMMARY:
Background:

Procalcitonin (PCT) is a biomarker that has been proposed as a helpful tool in inflammatory Clinique cases specially patient with pulmonary bacterienne infection .

Materials and methods the investigatore had retrospectively reviewed the electronic records and lists of all 582 COVID-19 patients admitted on the ICU of Hospital university Mohammed VI , Oujda. Between 01 juin 2020 and 31juanary 2021 , and analyzed the relation of PCT value and mortality at 30 days until we can defined a cut off Procalcitonine to use as a marker of severity and high mortality .

DETAILED DESCRIPTION:
Our objective is to assess the relationship between Procalcitonin and 30-day mortality in patients admitted to the resuscitation department of the Mohammed VI University Hospital Center, Oujda, Morocco, infected by the SARS COV 2 Virus .

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SARS COV2 infection needed admission in ICU .

Exclusion Criteria:

* patient under 15 ans

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: -582 patient with the SARS COV 2 virus, in the Resuscitation Service of the Mohammed VI University Hospital Center oujda, MAroc
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Procalcitonin is a marker of mortality | through study completion, an average of 8 mounths
  as a cutoff 0.5 ng/ml Procalcitonin could be used as mortality factors

CONTACTS AND LOCATIONS:
Locations (1):
- younes Oujidi, Berkane, Morocco

IPD SHARING:
Plan to Share IPD: No